CLINICAL TRIAL: NCT06162247
Title: Naples Federico II Intensive Cardiac Care Unit Registry (Naples FED2-ICCU Registry)
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giuseppe Gargiulo, Associate Professor, Federico II University
Other Study IDs: Naples FED2-ICCU Registry; CET Campania 3 86/2023 (Registry Identifier: Naples FED2-ICCU Registry)
Record Dates: First submitted 2023-11-18; First posted 2023-12-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Acute Cardiovascular Disease; Acute Coronary Syndrome; Acute Heart Failure; Cardiogenic Shock
MeSH Terms: conditions — Acute Coronary Syndrome; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This protocol proposes to prospectively evaluate current epidemiology, pharmacologic and invasive management and clinical outcomes of patients with acute cardiovascular diseases admitted at our ICCU.

DETAILED DESCRIPTION:
This study is designed as a single-center, investigator-initiated prospective observational study. Our ICCU is located at the Department of "Scienze Cardiovascolari, Diagnostica per Immagini, e Rete Tempo Dipendente delle Emergenze Cardiovascolari" of the Azienda Ospedaliera Universitaria Federico II. All scientific activities are performed in the Department of Advanced Biomedical Sciences of the University of Naples Federico II.

This is a prospective observational study which does not include pharmacologic or invasive treatments different from daily and guideline-directed management, but only collects data of patients for research purposes, therefore no specific treatments or procedures are included in this research protocol.

The Clinical Trial Unit at the University of Naples "Federico II" will oversee all study procedures and data management. The study data will be anonymized and managed using REDCap electronic data capture, which is hosted at the University of Naples "Federico II".

Once the patient is admitted to our ICCU, the informed consent will be signed and all data will be collected: demographic, clinical, procedural, therapeutic, and outcome data.

Clinical outcomes will be assessed in the in-hospital period, at 30 days, at 1-year and at the longest available follow-up (telephone or follow-up visit).

Main clinical outcomes will be adjudicated by an independent clinical events committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

1. Acute cardiovascular disease admitted at our ICCU
2. Age ≥18 years;
3. Written informed consent.

Exclusion Criteria:

1) Patients not providing consent to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with acute cardiovascular diseases admitted at our ICCU will be eligible for inclusion in the study, and only those not providing consent to data collection will be excluded.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2033-11-20 (Estimated); Study Completion 2033-11-20 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days, 1 year
  Number of patients with all-cause mortality
Cardiovascular mortality | 30 days, 1 year
  Number of patients with cardiovascular mortality
Myocardial infarction | 30 days, 1 year
  Number of patients with myocardial infarction
Stent thrombosis | 30 days, 1 year
  Number of patients with stent thrombosis
Stroke | 30 days, 1 year
  Number of patients with stroke
Heart Failure | 30 days, 1 year
  Number of patients with heart failure
Hospitalization for heart failure | 30 days, 1 year
  Number of patients with hospitalization for heart failure
Bleeding | 30 days, 1 year
  Number of patients with bleeding
Acute kidney injury | 30 days, 1 year
  Number of patients with acute kidney injury
Target vessel revascularization | 30 days, 1 year
  Number of patients with target vessel revascularization
Target lesion revascularization | 30 days, 1 year
  Number of patients with target lesion revascularization
Hospital length of stay | 0 to 30 days (or more depending on diration of hospitalization)
  Duration of hospitalization in days
Metrics of diuretic response and decongestion | 0 to 30 days (or more depending on diration of hospitalization)
  Diuresis quantification, weight loss, decongestion score, etc.
Poor neurologic outcomes | 30 days, 1 year
  Number of patients with poor neurologic outcomes
ICCU length of stay | 0 to 30 days (or more depending on diration of hospitalization)
  Duration of ICCU hospitalization in days
Metrics of need for mechanical circulatory support and vasopressors/inotropes | 0 to 30 days (or more depending on diration of hospitalization)
  Need for MCS, MCS type and duration; need for vasopressors/inotropes, vasopressors/inotropes types and duration
Quality of life | 30 days, 1 year
  Quality of life assessment by various scores or questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Gargiulo, MD, PhD, Principal Investigator — Department of Advanced Biomedical Sciences; Giovanni Esposito, MD, PhD, Study Chair — Department of Advanced Biomedical Sciences
Locations (1):
- Department of Advanced Biomedical Sciences, University Federico II of Naples, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2023 Oct 1;44(37):3627-3639. doi: 10.1093/eurheartj/ehad195. No abstract available. PMID 37622666
- [Background] Leonardi S, Montalto C, Carrara G, Casella G, Grosseto D, Galazzi M, Repetto A, Tua L, Portolan M, Ottani F, Galvani M, Gentile L, Cardelli LS, De Servi S, Antonelli A, De Ferrari GM, Visconti LO, Campo G; ACS Clinical Governance Programme Investigators. Clinical governance of patients with acute coronary syndromes. Eur Heart J Acute Cardiovasc Care. 2022 Nov 30;11(11):797-805. doi: 10.1093/ehjacc/zuac106. PMID 36124872
- [Background] Nadarajah R, Ludman P, Appelman Y, Brugaletta S, Budaj A, Bueno H, Huber K, Kunadian V, Leonardi S, Lettino M, Milasinovic D, Gale CP; NSTEMI Investigators. Cohort profile: the ESC EURObservational Research Programme Non-ST-segment elevation myocardial infraction (NSTEMI) Registry. Eur Heart J Qual Care Clin Outcomes. 2022 Dec 13;9(1):8-15. doi: 10.1093/ehjqcco/qcac067. PMID 36259751
- [Background] De Filippo O, D'Ascenzo F, Wanha W, Leonardi S, Raposeiras Roubin S, Fabris E, Truffa Giachet A, Huczek Z, Gaibazzi N, Ielasi A, Cortese B, Borin A, Nunez-Gil IJ, Ugo F, Marengo G, Bianco M, Barbieri L, Marchini F, Desperak P, Melendo-Viu M, Montalto C, Bruno F, Mancone M, Ferrandez-Escarabajal M, Morici N, Scaglione M, Tuttolomondo D, Gasior M, Mazurek M, Gallone G, Campo G, Wojakowski W, Abu Assi E, Sinagra G, de Ferrari GM. IncidenCe and predictOrs of heaRt fAiLure after acute coronarY Syndrome: The CORALYS registry. Int J Cardiol. 2023 Jan 1;370:35-42. doi: 10.1016/j.ijcard.2022.10.146. Epub 2022 Oct 25. PMID 36306949